CLINICAL TRIAL: NCT06677892
Title: Prospective, Non-interventional Study to Describe The Use of Maribavir and Its Effectiveness in Patients With Post-transplant Cytomegalovirus Infection/Disease in Line With Belgian Reimbursement Conditions (The MARIBEL Study)
Brief Title: A Study of Maribavir in Adults With Post-transplant Cytomegalovirus (CMV) Infection in Belgium
Acronym: MARIBEL
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4014
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with post-transplant CMV infection and/or disease that are refractory or intolerant to one or more prior therapies, who have undergone a solid organ transplant/ hematopoietic stem-cell transplantation (SOT/HSCT) and are treated with maribavir for the first time and in line with the Belgian reimbursement criteria, data will be collected and observed prospectively for up to 2 years.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
Cytomegalovirus (CMV) is a common virus that infects many people. It can cause serious illness in people with weak immune systems especially in those undergoing transplants. Maribavir is a medicine approved for treating CMV infection in adults after transplant.

The main aim of this study is to check the use of maribavir and learn how safe and effective in treating adults with CMV infection after transplant in Belgium in line with the Belgian reimbursement criteria.

During the study, a participant's data will be collected for 2 years. The study does not have fixed visits to the hospital, but it is recommended collect data from routine visits and contacts.

ELIGIBILITY:
Inclusion Criteria:

* Participant signed an informed consent form.
* Aged greater than or equal to (>=) 18 years at the time of consent.
* Received an HSCT/SOT.
* Diagnosed with CMV infection/disease any time after the HSCT/SOT date.
* Starting maribavir for the first time and in line with the Belgian reimbursement criteria.

Exclusion Criteria:

• Participant treated with maribavir before the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who had a CMV infection/disease after SOT/HSCT and who start maribavir, according to summary of product characteristics (SmPC) and in line with Belgian reimbursement criteria for maribavir will be included.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Effectiveness of Maribavir on CMV Viremia Clearance | Up to 16 weeks
  CMV viraemia clearance is defined as last CMV quantitative polymerase chain reaction (PCR) during maribavir treatment. Viral clearance plasma CMV DNA concentration below the lower limit of quantification (< LLOQ) less than [<] 137 international units per milliliters (IU/mL).
Duration of Treatment | From treatment start to discontinuation of maribavir (up to 16 weeks)
  Duration of treatment is defined as time from treatment start to discontinuation of maribavir.
Time to Viral Clearance | From treatment start to achievement of viral clearance (up to 2 years)
  Time to viral clearance is defined as time from treatment start to achievement of viral clearance.
Percentage of Participants With Drug Resistance | Up to 2 years
  Percentage of participants with drug resistance (UL97/UL27 genes) testing will be reported.
Number of Participants With Use of Maribavir in Daily Clinical Practice | Up to 16 weeks
Number of Participants Who Have Refractory CMV Infection With/Without Resistance, or Intolerance to a Previous CMV Treatment | Up to 16 weeks
  Refractory CMV infection with resistance is defined as viral genetic alteration that decreases susceptibility to one or more antiviral drugs.
Percentage of Participants With Recurrence After Maribavir Treatment | Up to 2 years
  Recurrence is defined as plasma CMV DNA concentration greater than or equal to (>=) LLOQ in 2 consecutive plasma samples, after achieving confirmed viremia clearance. Viremia clearance will be defined as plasma CMV DNA concentration below the lower limit of quantification (< LLOQ) that is <137 IU/mL.
Number of Participants With Treatment Related Adverse Events (AEs) | Up to 2 years
  The investigator is required to provide an assessment of the relationship of an AE to the studied drug(s), based on the consideration of all available information about the event, including temporal relationship to drug administration, recognized association with drug product/class, pharmacological plausibility, and alternative etiology (e.g., underlying illness, concurrent conditions, concomitant treatments). An related AE is defined as AE that follows a reasonable temporal sequence from administration of the medication, vaccine, or device (including the course after withdrawal of the medication), and for which a causal relationship is at least a reasonable possibility, i.e., the relationship cannot be ruled out, although factors other than the medication, vaccine, or device, such as underlying diseases, complications, concomitant drugs, and concurrent treatments, may also have contributed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- Belgium (9):
  - Hôpital Erasme, Anderlecht
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZA, Edegem
  - UZGent, Ghent
  - UZBrussel, Jette
  - UZLeuven, Leuven
  - CHU de Liège - site Sart Tilman, Liège
  - CHU UCL Namur - site Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/8db9463ef5b74455??page=1&idFilter=TAK-620-4014